CLINICAL TRIAL: NCT03360981
Title: Epicardial Fat Evaluation to Predict Clinical Outcomes in Patients Affected by Coronary Artery Disease and Treated by Coronary Artery Bypass Grafting: Diabetic vs. Non Diabetic Patients, and Incretin Therapy Effect; The EPI.FAT.IN Study
Brief Title: Epicardial Fat and Clinical Outcomes After Coronary Artery Bypass Grafting in Diabetics vs. Non Diabetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, MD, MSc, PhD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28.11.2017.1
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease | interventions — Incretins

STUDY DESIGN:
Intervention Model Description: arm 1 , diabetics treated by coronary artery bypass grafting (CABG), receiving epicardial tissue biopsy, and than treated by incretin therapy plus standard anti ischemic therapy..
  arm 2, diabetics, treated by coronary artery bypass grafting (CABG), receiving epicardial tissue biopsy, and than treated by standard hypoglycemic drug therapy plus standard anti ischemic therapy.
  arm 3, non diabetics, treated by coronary artery bypass grafting (CABG), receiving epicardial tissue biopsy, and than treated by standard anti ischemic therapy.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- diabetics incretin-users (arm 1) (Active Comparator): epicardial tissue biopsy, and than treated by incretin therapy plus standard anti ischemic therapy.
  Interventions: Drug: Incretins
- diabetics never-incretin-users (arm 2) (Placebo Comparator): epicardial tissue biopsy, and than treated by standard hypoglycemic drug therapy plus standard anti ischemic therapy.
  Interventions: Drug: Incretins
- non diabetics (arm 3) (No Intervention): non diabetics, treated by coronary artery bypass grafting (CABG), receiving epicardial tissue biopsy, and than treated by standard anti ischemic therapy.

INTERVENTIONS:
Drug: Incretins — after CABG, and epicardial tissue biopsy, patients will receive incretin therapy.
  Arms: diabetics incretin-users (arm 1); diabetics never-incretin-users (arm 2)

SUMMARY:
Cardiovascular disease (CVD) is a group of diseases including both the heart and blood vessels, thereby including coronary heart disease (CHD). To date, diabetics have a higher incidence and prevalence of multivessels CHD. Treatments in multivessels CHD in diabetics include full medical anti ischemic therapy, and revascularization therapy (Percutaneous coronary intervention (PCI) and/or Coronary artery bypass grafting (CABG)). Randomized trials comparing multivessel PCI to CABG have consistently demonstrated the superiority of CABG in reducing mortality, myocardial infarctions and need for repeat revascularizations. After the CABG treatment, diabetics vs. non-diabetics evidenced a worse prognosis, and an increased mortality. Numerous molecular, epigenetics (as microRNAs), and other metabolic risk factors may condition the worse prognosis in diabetics vs. non diabetics after CABG. In this context, an increased epicardial fat tissue thickness may be independently associated with the prevalence of diabetes, and diabetics have an higher epicardial fat tissue thickness, volumetry, and enhanced metabolism. Therefore, after CABG, lifestyle and medical improvements may lead to the reduction of epicardial fat thickness, extension, and metabolism in both non-diabetics, and diabetics, ameliorating the prognosis. At moment, epicardial tissue function in diabetics is not well investigated in literature, and no data has been reported about new hypoglycemic drugs, and its pleiotropic effects on diabetics after CABG. Indeed, our study hypothesis was that, epicardial fat tissue dimension, and metabolic activity may be related to a different expression of inflammatory, oxidative, and apoptotics molecules, and epigenetic effectors in diabetics vs. non-diabetics. Secondary, these effectors, and epicardial tissue dimension and activity, may be controlled, after CABG, by incretin treatment in diabetics. Therefore, incretin therapy may be associated to the reduction in epicardial fat tissue thickness, and extension, with down regulation of different inflammatory, oxidative and apoptotics molecules, and epigenetic effectors involved in epicardial fat metabolism. Moreover, in this study authors will evaluate in diabetics vs. non diabetics, and in diabetic incretin-users vs. never.-incretin-users, all cause mortality, cardiac mortality, and Major adverse cardiac events (MACE) after CABG in diabetics vs. non diabetics, and diabetic incretin-users (6 months of incretin therapy) vs. diabetic never-incretin-users. Authors will correlate these clinical endpoints to the study of the epicardial fat anatomy and metabolism before and after CABG, and to circulating inflammatory and pro-apoptotic markers, epigenetic effectors, and stem cells in diabetics vs. non diabetics, and diabetic incretin-users (6 months of incretin therapy) vs. diabetic never-incretin-users.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a group of diseases that include both the heart and blood vessels, thereby including coronary heart disease (CHD) and coronary artery disease (CAD), and acute coronary syndrome (ACS) among several other conditions. CHD causes about one-third of all deaths in people older than 35 years. Diabetes Mellitus (DM) is independently associated with a 2 to 4-fold increased mortality risk from heart disease, and with an increased mortality after myocardial infarction (MI), and worse overall prognosis with CAD. To date, DM patients have a higher incidence and prevalence of multivessels CAD. Treatments in multivessels CAD diabetics include full medical anti ischemic therapy (antiplatelets drugs, beta blockers, anti-remodelling drugs, anti-diabetic drugs etc), and revascularization therapy (Percutaneous coronary intervention (PCI) and/or Coronary artery bypass grafting (CABG)). Randomized trials comparing multivessel PCI to coronary artery bypass grafting (CABG) have consistently demonstrated the superiority of CABG in reducing mortality, myocardial infarctions and need for repeat revascularizations. After the CABG treatment, diabetics vs. non-diabetics evidenced a worse prognosis, and an increased mortality at follow up. The causes of the worse prognosis after CABG in diabetics are not well known, and under-investigated. Authors may speculate that, numerous molecular, epigenetics (as microRNAs), and other metabolic risk factors may condition the worse prognosis in diabetics vs. non diabetics after CABG. In this context, recently authors investigated the impact of epicardial adipose fat tissue dimension and metabolism on cardiovascular clinical outcomes. Intriguingly, an increased epicardial fat tissue thickness may be independently associated with the prevalence of diabetes. Consequently, diabetics have an higher epicardial fat tissue thickness, volumetry, and enhanced metabolism. Therefore, authors may speculate that, epicardial fat tissue may work as a metabolically active tissue, by a direct action on the heart, and by a cross talking with various metabolic derangements in the body leading to insulin resistance, atherosclerosis, metabolic syndrome, and cardiovascular disease. Moreover, after CABG, lifestyle and medical improvements may lead to the reduction of epicardial fat thickness, extension, and metabolism in both non-diabetics, and diabetics. Therefore, a part of the lifestyle modifications, also the hypoglycemic drugs therapy may lead to modification of epicardial fat tissue. However, authors may speculate that, the epicardial fat tissue thickness, volumetry, and metabolism, probably due to inflammatory and oxidative molecules activity, and epigenetic and anti-apoptotic pathways (as Sirtuins expression), may lead to a balance between epicardial fat tissue growth and/or reduction, and then all these pathways may be consequently involved in the prognosis of diabetics vs. non diabetics patients after CABG. At moment, all these pathways remain not well investigated in literature, and no data has been reported about new hypoglycemic drugs, and its pleiotropic effects on diabetics after CABG. Indeed, authors study hypothesis was that, epicardial fat tissue dimension, and metabolic activity may be related to a different expression of inflammatory, oxidative, and apoptotics molecules, and epigenetic effectors in diabetics vs. non-diabetics. Secondary, these effectors, and epicardial tissue dimension and activity, may be controlled, after CABG, by incretin treatment in diabetics. Moreover, higher epicardial fat tissue thickness, and tissue extension, may be associated with worse prognosis in diabetics after CABG. Secondary, in diabetics with better response to CABG, there may be a more important reduction of epicardial fat tissue tickness at follow up. This effect may be due to the control of different inflammatory, oxidative, and apoptotics molecules, and epigenetic effectors in diabetics undergoing CABG, and related to better clinical outcomes. Authors study hypothesis, is that incretin therapy may be associated to the reduction in epicardial fat tissue thickness, and extension. This effect in diabetics incretin-users vs. never-incretin-users may be due to the down regulation of different inflammatory, oxidative and apoptotics molecules, and epigenetic effectors involved in epicardial fat metabolism. Moreover, in this study authors will evaluate in diabetics vs. non diabetics, and in diabetic incretin-users vs. never.-incretin-users, all cause mortality, cardiac mortality, and Major adverse cardiac events (MACE) after CABG in diabetics vs. non diabetics, and diabetic incretin-users (6 months of incretin therapy) vs. diabetic never-incretin-users. Authors will correlate these clinical endpoints to the study of the epicardial fat anatomy and metabolism before and after CABG, and to the study of circulating inflammatory and pro-apoptotic markers, epigenetic effectors, and stem cells in diabetics vs. non diabetics, and diabetic incretin-users (6 months of incretin therapy) vs. diabetic never-incretin-users. A part of this, authors may speculate to recognize new cellular, molecular, and inflammatory processes, and epigenetic effectors epicardial fat derived related to these effects on clinical outcomes, and then used as specifical targets to improve clinical outcomes after CABG in diabetics.

ELIGIBILITY:
Inclusion Criteria:

* patients aged >18, <75, left ventricle ejection fraction (LVEF) >50%, multivessel coronary disease detected by coronarography, indication to receive a CABG, stable CAD. All diabetics and non diabetics.

Exclusion Criteria:

* acute myocardial infarction, heart failure, neoplastic disease, chronic diseases that may affect the inflammatory profile both systemic and epicardial (cancer, chronic intestinal inflammation, hepatitis, AIDS); life expectancy < 6 months, previous CABG and/or other open heart surgery intervention, acute coronary syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2019-08-20 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 12 months
  Authors will evaluate all cause of mortality in in diabetics vs. non diabetics, and in diabetics incretin-users vs. never-incretin-users by hospital discharge schedules, deaths registry, and during follow up visits.
cardiac mortality | 12 months
  Authors will evaluate cardiac mortality in in diabetics vs. non diabetics, and in diabetics incretin-users vs. never-incretin-users by hospital discharge schedules, deaths registry, and during follow up visits.
Major adverse cardiac events (MACE) | 12 months
  Authors will evaluate MACE in in diabetics vs. non diabetics, and in diabetics incretin-users vs. never-incretin-users by hospital discharge schedules, hospitalization schedules, and during follow up visits.

SECONDARY OUTCOMES:
molecular markers (Sirtuin 1, 6, etc) to predict study endpoints | 12 months
  Authors will evaluate sirtuin1, 6 etc in in diabetics vs. non diabetics, and in diabetics incretin-users vs. never-incretin-users by blood samples during hospitalization, and during follow up visits.
serum microRNAs and epicardial fat microRNAs, | 12 months
  Authors will evaluate serum microRNAs and epicardial fat microRNAs in diabetics vs. non diabetics, and in diabetics incretin-users vs. never-incretin-users by blood samples during hospitalization, and during follow up visits.clinical outcomes.
stem cells isolated in epicardial fat. | 12 months
  Authors will evaluate epicardial fat derived stem cells in diabetics vs. non diabetics, and in diabetics incretin-users vs. never-incretin-users by blood samples during hospitalization, and during follow up visits. Epicardial derived stem cells will be evaluated during CABG.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sardu C, D'Onofrio N, Torella M, Portoghese M, Loreni F, Mureddu S, Signoriello G, Scisciola L, Barbieri M, Rizzo MR, Galdiero M, De Feo M, Balestrieri ML, Paolisso G, Marfella R. Pericoronary fat inflammation and Major Adverse Cardiac Events (MACE) in prediabetic patients with acute myocardial infarction: effects of metformin. Cardiovasc Diabetol. 2019 Sep 30;18(1):126. doi: 10.1186/s12933-019-0931-0. PMID 31570103